CLINICAL TRIAL: NCT00825383
Title: Effect of Dietary Fiber on Glucose, Lipid, and Mineral Metabolism in Patients With Non Insulin Dependent Diabetes Mellitus
Brief Title: Effect of Dietary Fiber on Glucose & Lipids in Non Insulin Dependent Diabetes Mellitus (NIDDM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, Professor, Chairman Division Nutrition & Metabolic Diseases, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF498
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Non-Insulin-Dependent Diabetes Mellitus
Keywords: Diabetes; lipids; fiber
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): High Fiber Diet
  Interventions: Other: High Fiber and Moderate Fiber Diets
- 2 (Active Comparator): Moderate Fiber Diet
  Interventions: Other: High Fiber and Moderate Fiber Diets

INTERVENTIONS:
Other: High Fiber and Moderate Fiber Diets — Dietary
  Other Names: Dietary Fiber Study

SUMMARY:
Effect of Dietary Fiber on glucose, lipid, and mineral metabolism in patients with non insulin dependent diabetes mellitus.

DETAILED DESCRIPTION:
Two diets will be compared,a low fiber diet and a high fiber diet. These two diets will differ only in the content of total dietray fiber derived from natural food products. The diets will be identical in terms of total energy, percentage of total energy as proteins, fat and carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* NIDDM
* age 35 to 80 years
* stable oral hypoglycemic treatment for at least one month
* fasting triglycerides < 500 mg/dl

Exclusion Criteria:

* insulin dependent NIDDM
* insulin dependent diabetes
* hepatic disease
* significant hepatic dysfunction
* signifiacnt renal dysfunction
* presence of significant hematological, neurological, cardiovascular or gastrointestinal disorder, unless stable for past 6 months,
* serious intercurrent illness or anticipated major surgery
* female pregnant or likely to become pregnant
* chronic drug abuse, alcoholism or psychaitric disorder within the past 2 years
* treated with beta adrenergic blockers
* on lipid lowering drugs

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1993-01; Primary Completion 1995-12 (Actual); Study Completion 1995-12 (Actual)

PRIMARY OUTCOMES:
glucose and lipid metabolism | Baseline and during the last 5 days of each 6 week dietary phase

SECONDARY OUTCOMES:
calcium isotope absorption in the gastrointestinal tract, stool mineral content, 24 h urinary mineral concentration, and serum chemistry including mineral concentration. | Baseline and during the last 5 days of each 6 week dietary phase

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, Principal Investigator — UT Southwestern Medical Center at Dallas

REFERENCES:
- [Derived] Shah M, Chandalia M, Adams-Huet B, Brinkley LJ, Sakhaee K, Grundy SM, Garg A. Effect of a high-fiber diet compared with a moderate-fiber diet on calcium and other mineral balances in subjects with type 2 diabetes. Diabetes Care. 2009 Jun;32(6):990-5. doi: 10.2337/dc09-0126. Epub 2009 Mar 11. PMID 19279300